CLINICAL TRIAL: NCT04213001
Title: Diagnostic Contribution of Ultrasonography in Breast Cancer-Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Banu Dilek, Principal investigator, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DokuzEUBanuNihan
Record Dates: First submitted 2019-12-24; First posted 2019-12-30 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Lymphedema of Upper Arm
Keywords: Lymphedema; Circumferential measurements; ultrasonography
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- measure (Other): circumference measure, ultrasonographic measure
  Interventions: Diagnostic Test: ultrasonographic measurement

INTERVENTIONS:
Diagnostic Test: ultrasonographic measurement — ultrasonographic measurement- Subcutaneous ultrasound echogenicity (SEG) and Skin and subcutaneous thickness measurement

SUMMARY:
Breast cancer is the most common cancer in women. It is an important health problem that has been increasingly encountered in recent years. With advances in treatment, the survival time after breast cancer is prolonged, and as a result, many women face certain diseases during this period. One of these diseases, breast cancer-related lymphedema, is characterized by abnormal accumulation of protein-rich fluid in the interstitial tissue, which can occur at any time after breast cancer surgery or radiotherapy and is a major cause of morbidity.Early and accurate diagnosis of lymphedema is very important for effective treatment. In routine clinical practice there are various methods used to diagnose lymphedema such as history, physical examination and limb circumference. Circumferential measurement is based on the principle of circumference measurement at certain intervals (such as 4 cm, 5 cm, 10 cm) from certain anatomical reference points on the extremities. Volume calculation can also be made from a data obtained from circumferential measurements via a computer program. Circumferential and volume measurements are used in the diagnosis, severity of lymphedema and follow-up of treatment. Although it is the most commonly used method in practice, circumferential measurements and volume measurements alone can ignore changes in tissue structure and significant changes in the presence of latent lymphedema. At the same time, circumferential measurements are made at regular intervals and the difference between the healthy side and 2 cm or more is considered as lymphedema, which may neglect tissue and edema changes in areas not in the measuring area. Ultrasonography, which has been used in the measurement and evaluation of lymphedema in recent years, is a noninvasive economic method. Skin and subcutaneous distance in lymphedema can be measured by ultrasonography, and changes in tissue structure, fibrous tissue, adipose tissue and muscle tissue can be demonstrated. Fibrotic changes in lymphedema tissue play a key role in progression. Subcutaneous ultrasound echogenicity (SEG), which is thought to be a measure of lymphedema severity in extremities, was determined as stages 0, 1 and 2. According to this; Stage 0: No increase in echogenicity in the subcutaneous layer. That is, the subcutaneous fat layer is observed as black. Stage 1: Diffuse increase in echogenicity, but identifiable horizontal or oblique-focused echogenic lines caused by bundles of connective tissue may be seen. In this study, the investigators aimed to determine the correlation between circumferential measurements and skin and subcutaneous tissue ultrasonography in breast cancer-related lymphedema patients.The primer aim of this study is to investigate the correlation between circumferential measurements and ultrasonographic measurements in breast cancer-related lymphedema. The secondary aim is to investigate the relationship among the changes in subcutaneous tissue structure (subcutaneous ultrasound echogenicity degree-SEG) and lymphedema severity in breast cancer-related lymphedema.

DETAILED DESCRIPTION:
Patients with unilateral breast cancer-related lymphedema will be included in the study. The circumferences will be measured with a measuring tape from wrist ulnar styloid to axilla at 4 cm intervals. The point where the difference between the upper extremities was highest and the control point with no difference in the lower extremities will be marked. Ultrasonographic skin and subcutaneous thickness measurements will be performed from 4 quadrants; volar medial-lateral and dorsal medial-lateral sides of the extremity, with the probe placed transverse and perpendicular to the skin at the marked points.

The severity of lymphedema was graded ultrasonographically according to the SEG scale. (Stage 0: No increase in echogenicity in the subcutaneous layer. That is, subcutaneous fat is observed as black. Stage 1: Diffuse increase in echogenicity, but identifiable horizontal or oblique-oriented echogenic lines caused by bundles of connective tissue can be seen. Stage 2: A widespread increase in echogenicity echogenic lines cannot be identified.) Spearman test was used for correlations and Receiver Operating Characteristics (ROC) curve analysis was used to estimate the diagnostic accuracy. Sensitivity and specificity were calculated using a statistically significant threshold. Differences between ultrasonographic measurements between control points in lower extremities were compared with Wilcoxon test.

The minimum number of patients to be included in the study, according to the G-Power program, effect size d = 0.5, alpha-α = 0.05 and power 0.80 was calculated to be at least 34.

ELIGIBILITY:
Inclusion Criteria:

1. To be diagnosed with breast cancer-related unilateral lymphedema
2. Being over 18 years old
3. Having a female gender

Exclusion Criteria:

1. Bilateral breast cancer
2. Existing upper extremity infection
3. Lymphangitis
4. Refusal to participate in the study
5. Presence of edema in lower extremity

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
ultrasonographic measurement | baseline
  - Subcutaneous ultrasound echogenicity (SEG) and Skin and subcutaneous thickness measurement

CONTACTS AND LOCATIONS:
Overall Officials: Banu Dilek, Study Director — Dokuz Eylul University
Locations (1):
- Dokuz eylul university, Izmir, Inciralti, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Erdinc Gunduz N, Dilek B, Sahin E, Ellidokuz H, Akalin E. Diagnostic Contribution of Ultrasonography in Breast Cancer-Related Lymphedema. Lymphat Res Biol. 2021 Dec;19(6):517-523. doi: 10.1089/lrb.2020.0068. Epub 2021 Feb 18. PMID 33601960